CLINICAL TRIAL: NCT03702751
Title: Comparative Study Between Skin Adhesive Steristrips and Subcuticular Suture for Episiotomy Skin Repair in Primigravid Obese Women: A Randomized Controlled Trial
Brief Title: Steristrips Adhesive Tape Versus Subcuticular Suture for Episiotomy Repair in Primigravid Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: episiotomy
Record Dates: First submitted 2018-10-06; First posted 2018-10-11 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Episiotomy Wound
MeSH Terms: interventions — Surgical Tape

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesive tape (Experimental): will be subjected to skin repair after episiotomy with skin adhesive tape.
  Interventions: Procedure: Adhesive tape
- Continuous subcuticular skin suturing (Active Comparator): will be subjected to skin repair after episiotomy with the currently traditional method for episiotomy repair by continuous absorbable subcuticular suture.
  Interventions: Procedure: Continuous subcuticular skin suturing

INTERVENTIONS:
Procedure: Adhesive tape — will be subjected to skin repair after episiotomy with skin adhesive tape.
  Arms: Adhesive tape
Procedure: Continuous subcuticular skin suturing — will be subjected to skin repair after episiotomy with the currently traditional method for episiotomy repair by continuous absorbable subcuticular suture.
  Arms: Continuous subcuticular skin suturing

SUMMARY:
This study will be done to question the superiority of using skin adhesive tape (® Steri-Strip) closure in wound pain and healing over the traditional running absorbable subcuticular suture technique in perineal repair after episiotomy in obese primiparous women..

DETAILED DESCRIPTION:
Episiotomy is the most common operating procedure that most obstetricians will perform in their lifetime. Because it is so common and considered minor surgery, teaching students or interns the principles and techniques usually is left to the most junior of residents

The optimal method for episiotomy and perineal trauma repair following childbirth remains open to debate and a great cause of concern to doctors, midwives, and the public

Apparently, the ideal method for perineal repair should be quick, painless, easy to perform and preferably, without an increase in pain and dyspareunia during the puerperium

This study will be commenced to question the advantage of using skin adhesive tape (® Steri-Strip) closure in wound pain and healing over the traditional running absorbable subcuticular suture technique in perineal repair after episiotomy in obese primiparous women.

ELIGIBILITY:
Inclusion Criteria:

* primigravidae 18 years or older.
* Spontaneous not induced full term normal not instrumental vaginal delivery with mediolateral episiotomy.
* First and 2nd-degree perineal tear.
* BMI≥30

Exclusion Criteria:

* • patients who had an instrumental delivery.

  * 3rd and fourth-degree perineal tears.
  * those with local infectious lesions in the area to be repaired.
  * preexisting medical disorders as diabetes mellitus, severe pulmonary disease and collagen disease.
  * Immunosuppressive treatment.
  * known hypersensitivity to adhesive tape or materials.
  * Maternal unwillingness to undergo randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Severity of pain 6h postoperatively | 6 hours after the procedure
  the patient will report her pain by placing a line perpendicular to the VAS line at the point that represents their pain intensity.VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain.
Severity of pain 12 hours postpartum | 12 hours after the procedure
  the patient will report her pain by placing a line perpendicular to the VAS line at the point that represents their pain intensity. VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain.

SECONDARY OUTCOMES:
wound healing | 7-10 days after delivery
  During the second visit 7-10 days after delivery; wound healing will be evaluated and recorded by Redness, Edema, Ecchymosis, Drainage, Approximation (REEDA), data may be collected by home visits for those may not be able to come back for the second visit.
Severity of pain 10 days postpartum | 10 days after procedure
  pain experience will be evaluated by visual analog scale
timing of procedure | During the procedure
  timing of both procedures will be recorded and documented
Severity of pain immediately after episiotomy repair | immediately after the procedure
  pain experience will be evaluated immediately after the procedure by the visual analog scale(VAS). VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Ashour, Giza, Egypt